CLINICAL TRIAL: NCT00940316
Title: A Randomized Phase II Study of Dual Epidermal Growth Factor Receptor Inhibition With Erlotinib and Panitumumab With or Without Irinotecan as Second Line Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: Dual Epidermal Growth Factor Receptor Inhibition With Erlotinib and Panitumumab With or Without Chemotherapy for Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry); Amgen (Industry)
Responsible Party: Principal Investigator, Al Benson, Al Benson, MD, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 07I4; STU00004101 (Other: Northwestern University IRB); OSI 4263s (Other: OSI Pharmaceuticals, Inc)
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Panitumumab; Erlotinib Hydrochloride; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Erlotinib + Panitumumab + Irinotecan (Experimental): Patients receive oral erlotinib hydrochloride once daily on days 1-14, panitumumab IV over 30-90 minutes on day 1, and irinotecan hydrochloride IV over 90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: panitumumab; Drug: erlotinib hydrochloride; Drug: irinotecan hydrochloride
- Arm B: Erlotinib + Panitumumab (Experimental): Patients receive oral erlotinib hydrochloride once daily on days 1-14 and panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients receive irinotecan hydrochloride as in arm A.
  Interventions: Biological: panitumumab; Drug: erlotinib hydrochloride; Drug: irinotecan hydrochloride
- Arm C: Erlotinib + Panitumumab (Experimental): Patients receive erlotinib hydrochloride and panitumumab as in arm B.
  Interventions: Biological: panitumumab; Drug: erlotinib hydrochloride

INTERVENTIONS:
Biological: panitumumab — Given intravenously 6mg/kg every 2 weeks
  Other Names: Vectibix
Drug: erlotinib hydrochloride — Given orally 150mg daily
  Other Names: Tarceva
Drug: irinotecan hydrochloride — Given intravenously 120mg/m2 for 6/6 genotype and 60mg/m2 for 6/7 genotype
  Other Names: Camptosar; CPT-11
  Arms: Arm A: Erlotinib + Panitumumab + Irinotecan; Arm B: Erlotinib + Panitumumab

SUMMARY:
RATIONALE: Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Panitumumab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether erlotinib hydrochloride given together with panitumumab is more effective with or without irinotecan in treating patients with metastatic colorectal cancer.

PURPOSE: This randomized phase II trial is studying giving erlotinib hydrochloride together with panitumumab to see how well it works with or without irinotecan hydrochloride as second-line therapy in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with metastatic colorectal cancer treated with erlotinib hydrochloride and panitumumab with versus without irinotecan hydrochloride as second-line therapy .

Secondary

* Determine time to disease progression and time to treatment failure in patients treated with these regimens.
* Determine the safety of these regimens in these patients.
* Determine the effect of these regimens on downstream targets of EGFR in skin rash associated with pharmacologic EGFR inhibition (exploratory).
* Determine the association between KRAS mutations and response to EGFR inhibition (exploratory).

OUTLINE: This is a multicenter study. Patients are stratified according to wild-type Kras tumors ( 6/6 UGT1A1 vs 6/7 UGT1A1), and are randomized to 1 of 2 treatment arms. Patients with wild-type Kras tumor 7/7 UGT1A1 receive treatment in arm III.

* Arm I: Patients receive oral erlotinib hydrochloride once daily on days 1-14, panitumumab IV over 30-90 minutes on day 1, and irinotecan hydrochloride IV over 90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral erlotinib hydrochloride once daily on days 1-14 and panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients receive irinotecan hydrochloride as in arm I.
* Arm III: Patients receive erlotinib hydrochloride and panitumumab as in arm II. Skin biopsies and blood samples may be collected for further analysis.

After completion of study therapy, patients are followed every 6 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Metastatic disease

    * Biopsy of either the primary cancer or metastatic site required
  * Tumor expressing wild-type Kras mutations
* Progressive disease within 3 months after treatment with first-line fluorouracil (5-FU) and oxaliplatin-based chemotherapy OR evidence of metastatic disease within 6 months of completing adjuvant therapy with 5-FU and oxaliplatin
* Measurable disease defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques OR as ≥ 10 mm with spiral CT scan

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 6 months
* ANC > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Creatinine < 1.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN (or < 2 mg/dL)
* AST and/or ALT < 3 times ULN (< 5 times ULN with liver metastases)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent malignancy requiring therapy except minor surgery for non-melanoma skin cancer removal
* No interstitial lung disease with symptoms (e.g., dyspnea or cough) including any of the following significant conditions:

  * Parenchymal lung disease
  * Metastatic disease
  * Pulmonary infections

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior EGFR inhibitors, irinotecan hydrochloride, or other second-line chemotherapy regimens
* More than 4 weeks since prior radiotherapy
* No other concurrent investigational agents
* No other concurrent anticancer treatment modalities (e.g., radiotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01-18 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al Benson, MD, Principal Investigator — Northwestern University
Locations (10):
- United States (10):
  - Cancer Care & Hematology Specialists of Chicagoland, Arlington Heights, Illinois
  - Northwestern University, Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Hematology/Oncology Associates, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Hope Cancer Center, Terre Haute, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Virtua Memorial (Regional Cancer Care Associates of Mount Holly), Mount Holly, New Jersey
  - Mercy Clinic Oncology and Hematology, Oklahoma City, Oklahoma
  - The Jones Clinic, Germantown, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on July 9, 2009 with an accrual goal of up to 96 patients. The study was designed to enroll 13 patients on each arm and do an interim efficacy assessment. Accrual was suspended on March 31 2015 fand closed permanently on April 13, 2015 with 28 patients enrolled on the study.
Pre-assignment Details: Subjects with either 6/6 UGT1A1 genotype or 6/7 UGT1A1 genotype will be randomized into either Arm A and Arm B. Subjects with 7/7 UGT1A1 genotype enrolled in Arm C.
Period: Reached First Response at 8 Weeks
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab
Started | 13 | 13 | 2
Completed | 10 | 9 | 2
Not Completed | 3 | 4 | 0
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Progressive disease | 1 | 3 | 0
Period: Moved on to be Treated Cycle 5
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab
Started | 10 | 9 | 2
Completed | 8 | 9 | 2
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Period: Treated After Cycle 5
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab
Started | 8 | 9 | 2
Completed | 8 | 8 | 1
Not Completed | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Progressive disease | 0 | 1 | 0
Period: Crossed Over to Arm A After Progression
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab
Started (Patients on Arm B that progressed were able to cross over and be treated on arm A if still eligible.) | 0 | 3 | 0
Treated for Cycle One | 0 | 3 | 0
Completed | 0 | 3 | 0
Not Completed | 0 | 0 | 0
Period: Follow up Every 3 Months
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab
Started (All patients that receive treatment on the study go into follow up at treatment completion.) | 13 | 13 | 2
Completed | 13 | 13 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab | Total
Number analyzed (Participants) | 13 | 13 | 2 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 2 | 19
  >=65 years | 5 | 4 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 0 | 11
  Male | 7 | 8 | 2 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 5
  Not Hispanic or Latino | 10 | 11 | 2 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 12 | 12 | 1 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 2 | 28
UGT1A1 genotyping 6/6 [Count of Participants; unit: Participants] | 9 | 7 | 0 | 16
UGT1A1 genotyping 6/7 [Count of Participants; unit: Participants] | 4 | 6 | 0 | 10
UGT1A1 genotyping 7/7 [Count of Participants; unit: Participants] | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate Based on Complete Response (CR)+ Partial Response (PR) + Stable Disease (SD)
Description: Tumor response rate will be measured by CT scan of the chest and CT scan or MRI scan of abdomen and pelvis every 8 weeks until disease progression response rate will be measured per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions evaluated using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions.
  Complete Response (CR): Disappearance of all target lesions.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD)of target lesions, taking as reference the baseline sum LD.
  Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions,taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: At baseline and every 8 weeks during treatment until progressive disease for maximum of 51 cycles where 1 cycle = 2 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Erlotinib + Panitumumab + Irinotecan: Arm A - Patients receive oral erlotinib hydrochloride once daily on days 1-14, panitumumab IV over 30-90 minutes on day 1, and irinotecan hydrochloride IV over 90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
  panitumumab: Given intravenously 6mg/kg every 2 weeks
  erlotinib hydrochloride: Given orally 150mg daily
  Irinotecan hydrochloride: Given intravenously 120mg/m2 every 2 weeks
- Arm B: Erlotinib + Panitumumab: Arm B - Patients receive oral erlotinib hydrochloride once daily on days 1-14 and panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients receive irinotecan hydrochloride as in arm A.
  panitumumab: Given intravenously 6mg/kg every 2 weeks
  erlotinib hydrochloride: Given orally 150mg daily
- Arm C: Erlotinib + Panitumumab: Arm C - Patients receive erlotinib hydrochloride and panitumumab as in arm B.
  panitumumab: Given intravenously 6mg/kg every 2 weeks
  erlotinib hydrochloride: Given orally 150mg daily
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab
Number analyzed (Participants) | 13 | 13 | 2
Participants
  Complete Response | 0 | 1 | 0
  Partial Response | 4 | 3 | 0
  Stable disease | 6 | 3 | 2

2. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression will be measured by CT scan of the chest and CT scan or MRI scan of abdomen and pelvis every 8 weeks until disease progression . Time to disease progression will be defined as the time elapsed from the day of 1st study drug administration to the day disease progression is documented or death occurs and will .
  Progressive Disease will be defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) : At least a 20% increase in the sum of the longest diameter (LD) of target lesions,taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: At baseline and every 8 weeks during treatment until disease progression and for a maximum of 51 cycles where 1 cycle = 2 weeks
Population: All patient data analyzed reported together regardless of arm allocation. Data not collected and analyzed for this outcome measure.
Groups:
- Arm A + Arm B + Arm C: Arm A - Patients receive oral erlotinib hydrochloride once daily on days 1-14, panitumumab IV over 30-90 minutes on day 1, and irinotecan hydrochloride IV over 90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Arm B - Patients receive oral erlotinib hydrochloride once daily on days 1-14 and panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients receive irinotecan hydrochloride as in arm A.
  Arm C - Patients receive erlotinib hydrochloride and panitumumab as in arm B.
  panitumumab: Given intravenously 6mg/kg every 2 weeks
  erlotinib hydrochloride: Given orally 150mg daily
  Irinotecan hydrochloride: Given intravenously 120mg/m2 every 2 weeks
Arm/Group | Arm A + Arm B + Arm C
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure will be measured as the time elapsed from the day of first study drug administration to the date a subject stops all study drugs for any reason.
Time Frame: From first day of study drug treatment until the date of stopping all study drugs for any reason for a maximum of 51 cycles where 1 cycle=2weeks
Population: Data was not collected and analyzed for this outcome measure
Arm/Group | Arm A + Arm B + Arm C
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicity of the Combination of Study Drugs
Description: Data on the toxicity of the combination of study drugs is assessed by laboratory blood draws done on day 1 of every treatment cycle and by patient report while on study treatment and up to 30 days after the last treatment. Grade 3 and grade 4 adverse events (AE) where the relationship between the AE and at least one of the study drugs were considered to be definite, probable or possible, were collected using National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0). AEs are graded as:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: Day 1 of every 2 week treatment cycle while on study treatment and 30 days after the last treatment for a maximum of 51 cycles.
Measure: Number; unit: participants
Groups:
- Arm B Cross Over - Erlotinib + Panitumumab + Irinotecan: Patients receive oral erlotinib hydrochloride once daily on days 1-14 and panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients receive irinotecan hydrochloride as in arm A.
  panitumumab: Given intravenously 6mg/kg every 2 weeks
  erlotinib hydrochloride: Given orally 150mg daily
  irinotecan hydrochloride: Given intravenously 120mg/m2 for 6/6 genotype and 60mg/m2 for 6/7 genotype
  After progression patients cross over to Arm A and Irinotecan is added. irinotecan hydrochloride IV over 90 minutes on day 1 or a 14 day cycle.
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab | Arm B Cross Over - Erlotinib + Panitumumab + Irinotecan
Number analyzed (Participants) | 13 | 10 | 2 | 3
participants
  Hemoglobin decrease | 3 | 1 | 0 | 0
  Leukocyte decrease | 7 | 0 | 1 | 0
  Lymphopenia | 1 | 0 | 0 | 0
  Neutrophil decrease | 7 | 0 | 1 | 0
  Fatigue | 1 | 1 | 1 | 0
  Dry skin | 1 | 0 | 0 | 0
  Rash/desquamation | 0 | 0 | 1 | 0
  Rash: Hand-foot skin reaction | 4 | 7 | 2 | 0
  Anorexia | 1 | 0 | 0 | 0
  Diarrhea | 6 | 0 | 1 | 0
  Nausea | 1 | 0 | 1 | 0
  Infection | 1 | 0 | 0 | 0
  Alkaline phosphatase decrease | 0 | 2 | 0 | 0
  Magnesium decrease | 5 | 4 | 1 | 0
  Phosphate decrease | 2 | 1 | 3 | 0
  Sodium decrease | 1 | 0 | 0 | 0
  Syncope/fainting | 1 | 0 | 0 | 0
  Pruritus/itching | 0 | 1 | 0 | 0

5. Secondary Outcome: Effect on Downstream Targets of Epidermal Growth Factor Receptor (EGFR) in Skin Rash Associated With Pharmacologic EGFR Inhibition
Description: Effect on downstream targets of EGFR in skin rash associated with pharmacologic EGFR inhibition. Skin biopsies will be performed at baseline (before the first days of treatment) and and at a time-point reflecting maximum rash intensity determined by a dermatologist.
Time Frame: At baseline and at a time-point reflecting maximum rash intensity during treatment, at a maximum of 51 cycles.
Population: All patient data analyzed reported together regardless of arm allocation.This outcome measure was based on optional biopsies that patients were required to consent to. Data was not collected or analyzed for this outcome measure.
Arm/Group | Arm A + Arm B + Arm C
Number analyzed (Participants) | 0

6. Post Hoc Outcome: Median Overall Survival
Description: Median Overall Survival (OS) is measured from treatment initiation until death due to any cause.
Time Frame: From the time of first treatment to death
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm A: Erlotinib + Panitumumab + Irinotecan: Arm A - Patients receive oral erlotinib hydrochloride once daily on days 1-14, panitumumab IV over 30-90 minutes on day 1, and irinotecan hydrochloride IV over 90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Arm B - Patients receive oral erlotinib hydrochloride once daily on days 1-14 and panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients receive irinotecan hydrochloride as in arm A.
  Arm C - Patients receive erlotinib hydrochloride and panitumumab as in arm B.
  panitumumab: Given intravenously 6mg/kg every 2 weeks
  erlotinib hydrochloride: Given orally 150mg daily
  Irinotecan hydrochloride: Given intravenously 120mg/m2 every 2 weeks
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab
Number analyzed (Participants) | 13 | 13 | 2
Months | 12.6 [4.8 to 19.4] | 8.6 [3.1 to 30.1] | 2.4 [NA to NA] — Sample size to small to calculate confidence interval

7. Post Hoc Outcome: Progression Free Survival (PFS)
Description: Progression free survival will be measured every 8 weeks during treatment by CT or MRI scans. Progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST).
  Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm B: Erlotinib + Panitumumab: Arm B - Patients receive oral erlotinib hydrochloride once daily on days 1-14 and panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients receive irinotecan hydrochloride as in arm A.
  Arm C - Patients receive erlotinib hydrochloride and panitumumab as in arm B.
  panitumumab: Given intravenously 6mg/kg every 2 weeks
  erlotinib hydrochloride: Given orally 150mg daily
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab
Number analyzed (Participants) | 12 | 13 | 2
Months | 4.6 [1.4 to 8.2] | 3.8 [1.5 to 5.9] | 2.4 [NA to NA] — Sample size too small to calculate confidence interval

ADVERSE EVENTS:
Time Frame: Adverse events (AE) for the study were collected over a 5 year period. AEs were collected for each patient whilst on treatment and for 30 days post last treatment for a maximum of up to 51 cycles (longest number of cycles any one patient received treatment)
Arm/Group | Arm A: Erlotinib + Panitumumab + Irinotecan | Arm B: Erlotinib + Panitumumab | Arm C: Erlotinib + Panitumumab | Arm B Cross Over - Erlotinib + Panitumumab + Irinotecan
All-Cause Mortality (participants affected / at risk) | 11/13 | 10/10 | 1/2 | 3/3
Serious Adverse Events (participants affected / at risk) | 3/13 | 4/10 | 1/2 | 1/3
Other Adverse Events (participants affected / at risk) | 13/13 | 10/10 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Erlotinib + Panitumumab + Irinotecan (N=13) | Arm B: Erlotinib + Panitumumab (N=10) | Arm C: Erlotinib + Panitumumab (N=2) | Arm B Cross Over - Erlotinib + Panitumumab + Irinotecan (N=3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Patient admitted for diarrhea but also had fatigue, neutropenic fever, nausea and vomiting during the hospital admission.
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient also experienced decreased white blood cell count
Death NOS- progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient also experienced drug induced pneumonitis during this hospital admission
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Partial Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Patient also experienced anemia and colonic fistula during this hospital admission.
Neutropenic fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient also experienced diarrhea, sepsis and rash during this hospital admission
Urinary Track infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Patient also experienced anemia during this hospital admission
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Patient also experiences esophagitis during this hospital admission
Altered mental status (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Erlotinib + Panitumumab + Irinotecan (N=13) | Arm B: Erlotinib + Panitumumab (N=10) | Arm C: Erlotinib + Panitumumab (N=2) | Arm B Cross Over - Erlotinib + Panitumumab + Irinotecan (N=3)
Hearing: patients without baseline audiogram and not enrolled in a monitoring (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hemoglobin (Anemia) (Blood and lymphatic system disorders) | 9 | 8 | 1 | 2
Neutrophils (neutropenia) (Blood and lymphatic system disorders) | 6 | 1 | 0 | 1
Leukocytes (total white blood cells) (Blood and lymphatic system disorders) | 9 | 1 | 0 | 1
lymphopenia (Blood and lymphatic system disorders) | 6 | 2 | 0 | 0
Platelets (thrombocytopenia) (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1
Elevated BUN (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hypertension (Cardiac disorders) | 4 | 2 | 0 | 0
Hypotension (Cardiac disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 8 | 4 | 0 | 1
Fever (General disorders) | 3 | 1 | 0 | 0
Insomnia (General disorders) | 1 | 0 | 0 | 0
Rigors (General disorders) | 2 | 0 | 0 | 0
Weight loss (General disorders) | 2 | 1 | 0 | 0
International Normalized Ratio of prothrombin time (INR) (Investigations) | 0 | 1 | 0 | 0
Cheilitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hair loss (alopecia) (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Acne/acneiform (Skin and subcutaneous tissue disorders) | 9 | 10 | 1 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Rash: Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Paronychia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Fungal infection beneath left breast (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pseudomonas (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Extensive growth of eyelashes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Scalp rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Face rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Glucose intolerance (Endocrine disorders) | 1 | 0 | 0 | 0
Anorexia (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 9 | 5 | 0 | 3
Distension/bloating of abdomen (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Mucositis/stomatitis (Gastrointestinal disorders) | 4 | 0 | 0 | 1
Heartburn (dyspepsia) (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 3 | 0 | 2
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Retal burning (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colon cancer with liver metastasis and likely bone metastasis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nosebleed (General disorders) | 1 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Infection in pelvis (with normal ANC or grade 1 or 2 neutrophils) (Infections and infestations) | 1 | 0 | 0 | 0
Infection in upper airway (with normal ANC or Grade 1 or 2 neutrophils) (Infections and infestations) | 0 | 1 | 0 | 0
Infection in abdomen (with normal ANC or Grade 1 or 2 neutrophils) (Infections and infestations) | 0 | 1 | 0 | 0
Infection in urinary tract (unknown ANC) (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (infection with grade 3 or 4 neutrophils) (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Cellulitis) (Infections and infestations) | 0 | 1 | 0 | 1
Ear infection (Infections and infestations) | 2 | 0 | 0 | 0
Pseudomonas Bactermia (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia coli (Infections and infestations) | 1 | 0 | 0 | 0
Edema - limb (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 8 | 3 | 0 | 2
Alkaline phosphatase increase (Metabolism and nutrition disorders) | 5 | 6 | 2 | 2
ALT increase (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 5 | 2 | 1 | 2
AST increase (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 8 | 6 | 2 | 3
Bilirubin increase (hyperbilirubinemia) (Metabolism and nutrition disorders) | 6 | 4 | 1 | 2
Creatinine increase (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Creatine phosphokinase (CPK) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Calcium, serum high (hypercalcemia) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Calcium, serum low (hypocalcemia) (Metabolism and nutrition disorders) | 7 | 2 | 0 | 2
Glucose, serum high (hyperglycemia) (Metabolism and nutrition disorders) | 7 | 4 | 0 | 0
Magnesium, serum low (hypomagnesemia) (Metabolism and nutrition disorders) | 10 | 10 | 2 | 3
Phosphate, serum low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 | 3 | 0 | 3
Potassium, serum high (hyperkalemia) (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Potassium, serum low (hypokalemia) (Metabolism and nutrition disorders) | 10 | 6 | 1 | 3
Sodium, se high (hypernatremia) (Metabolism and nutrition disorders) | 3 | 3 | 0 | 1
Sodium, serum low (hyponatremia) (Metabolism and nutrition disorders) | 4 | 3 | 2 | 1
Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0
Confusion (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 1 | 1
Depression (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Fainting (syncope episode) (Nervous system disorders) | 1 | 0 | 0 | 0
Muscle weakness generalized (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck stiffness (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Abdomen pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Extremity/limb pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rectum pain (General disorders) | 1 | 0 | 0 | 0
Flank pain (General disorders) | 0 | 1 | 0 | 0
Pain NOS (General disorders) | 1 | 0 | 0 | 0
Pain in throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 1
Eye lesion (Eye disorders) | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0
Meibomian gland dysfunction (Eye disorders) | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0
Cloudy vision (Eye disorders) | 1 | 0 | 0 | 0
Eythema/conjunctive (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Urine color change (Renal and urinary disorders) | 1 | 0 | 0 | 0
Decreased GFR (Renal and urinary disorders) | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Oral dysesthesia (General disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Sponsor did not renew contract and only 28 patients of the anticipated 96 were enrolled and treated on the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes